CLINICAL TRIAL: NCT05926986
Title: Investigation of Cognitive Functions in Patients With Fibromyalgia Syndrome
Brief Title: Cognitive Functions in Patients With Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Firat University, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-21
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; cognitive functions; exercise
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Aerobic exercise will be performed to all participants for a single session. Maximum heart rate was calculated for each subject (220 - age) and a heart rate monitor (Polar FT 100, China) will be used to follow subjects' heart rate during aerobic exercise. Additionally, pilates exercises will be performed three days in a week. Treatment will continue an hour in per session for 8 weeks.
  Interventions: Other: Exercise
- Control group (Experimental): No additional treatment will be practiced to the control group.
  Interventions: Other: control

INTERVENTIONS:
Other: Exercise — Aerobic exercise will be performed to all participants for a single session. Maximum heart rate was calculated for each subject (220 - age) and a heart rate monitor (Polar FT 100, China) will be used to follow subjects' heart rate during aerobic exercise. Additionally, pilates exercises will be performed three days in a week. Treatment will continue an hour in per session for 8 weeks.
  Arms: Study group
Other: control — No additional treatment will be practiced to the control group.
  Arms: Control group

SUMMARY:
Accumulating research with human adults suggests that a single session of physical exercise ameliorates different aspects of cognitive function immediately after the end of the exercise period, regardless of fitness level. It has now been more clearly demonstrated that the effect of physical exercise on cognitive performance depends both on the intensity and the duration of the exercise. Fibromyalgia (FM) is a complex clinical syndrome characterized by chronic widespread musculoskeletal pain, sleep disturbances, morning stiffness, fatigue, anxiety, and depressive symptoms. The aim of the study is to investigate the effects of exercise on cognitive functions in patients with FM.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a complex clinical syndrome characterized by chronic widespread musculoskeletal pain, sleep disturbances, morning stiffness, fatigue, anxiety, and depressive symptoms. Its etiology is not known, and several aspects of its pathogenesis are being investigated, shedding some light on the possible physiopathologic mechanisms involved in this process.The high prevalence of cognitive dysfunction reported among patients with fibromyalgia (50-80%), and the fact that memory and concentration problems can be very disruptive for patients, makes central to find strategies aiming at improving cognition in this population. Among non-pharmacological treatment options, enhancing physical fitness (mainly through physical exercise) or decreasing body fatness are becoming increasingly popular for improving the fibromyalgia-related symptomatology (including cognitive functioning) and quality of life. Accumulating research with human adults suggests that a single session of physical exercise ameliorates different aspects of cognitive function immediately after the end of the exercise period, regardless of fitness level. It has now been more clearly demonstrated that the effect of physical exercise on cognitive performance depends both on the intensity and the duration of the exercise.The aim of the study is to investigate the effects of exercise on cognitive functions in patients with FM.

Methods: Forty patients diagnosed with FMS according to the 2016 ACR criteria will be included in the study. While patients aged 18-65 whose medical treatment has not changed in the last three months will be included; Patients with pregnancy or malignancy diagnosis, systemic inflammatory rheumatic disease, neurological, orthopedic or congenital problems that prevent physical activity, and regular exercise habits will be excluded from the study. Patients who meet the criteria and agree to participate in the study will be divided into two groups. Routine treatments will be continued without any application to the control group. In the study group, aerobic and pilates exercises combined (30 minutes aerobic exercise to be performed on the treadmill at 60% of the maximum heart rate for 30 minutes, pilates exercises for 30 minutes) in Fırat University Physical Therapy and Rehabilitation Treatment Units, each session lasting approximately one hour, three days a week. ) will be applied. Treatment will continue for eight weeks. The patients participating in the study will be evaluated in their first sessions before starting the treatment and at the end of the treatment (in the eighth week). Stroop Test, verbal fluency test and Beck Depression Inventory will be applied to evaluate cognitive and psychosocial functions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were aged between 18-65 years,
* Patients who got diagnosed with Fibromyalgia Syndrome

Exclusion Criteria:

* Patients who had regular exercise habits, malignancy, pregnancy, incorporation,
* Patients who had changes of medical treatment in last 3 months
* Patients who diagnosed with Osteoarthritis for lower extremity
* Patients who had cardiac symptoms according to New York Heart Association
* Patients who had dysfunction that can prevent physical activity

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-10-20 (Estimated)

PRIMARY OUTCOMES:
The Stroop Color and Word Test | 2 minutes
  The Stroop Color and Word Test (SCWT) is a neuropsychological test extensively used for both experimental and clinical purposes. It assesses the ability to inhibit cognitive interference, which occurs when the processing of a stimulus feature affects the simultaneous processing of another attribute of the same stimulus

SECONDARY OUTCOMES:
Beck Depression Inventory | 1 minute
  Turkish version of Beck Depression Inventory (BDI) will be used to determine the depression levels of subjects. It consists of 21 items regarding pessimism, guilt, sleep, appetite and fatigue and each item is scored between 0 and 3. Higher scores shows the severity of depression.Score > 18 of BDI was considered as a cut-off value for depression.
Verbal Fluency test | 2 minutes
  The Verbal Fluency Test consists of lexical and semantic fluency tests. Sustained attention and vocabulary skill scanning ability are measured. The patient is asked to say as many words containing given letters (K, A, S) as possible in a minute, for word fluency. In category fluency, the patient is asked to say as many animal names as he or she can. The total number of words found is included to the scores.

CONTACTS AND LOCATIONS:
Overall Officials: Songül Bağlan Yentür, Principal Investigator — Firat University
Locations (1):
- Songül Bağlan Yentür, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Exercise therapy for fibromyalgia — http://pubmed.ncbi.nlm.nih.gov/21725900/
- See also: Exercise, fibromyalgia, and fibrofog: a pilot study — http://pubmed.ncbi.nlm.nih.gov/19420402/